CLINICAL TRIAL: NCT02599441
Title: Comparison of a Novel Weight Bearing Cone-beam Computed Tomography (CT) Scan to Gravity Stress X-ray for Determining Instability of Supination-external Rotation Type Ankle Fractures
Brief Title: Computed Tomography for Evaluating Supination-external Rotation Type Ankle Fractures
Status: Completed | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, John Marzo, Associate Professor of Clinical Orthopaedics, State University of New York at Buffalo
Other Study IDs: 733368-1
Record Dates: First submitted 2015-11-04; First posted 2015-11-06 (Estimated); Results first posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Supination-external Rotation Ankle Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ankle fracture cases

SUMMARY:
To compare measures of ankle stability from an investigational cone beam computed tomography scanner to gravity stress X-ray in patients who have unstable supination-external rotation ankle fractures.

ELIGIBILITY:
Inclusion Criteria:

* willing & able to provide written informed consent
* at least 18 years-old
* have medial clear space measuring less than 5 mm with clinical suspicion of instability and would normally require a gravity stress X-ray

Exclusion Criteria:

* pregnant (females)
* prisoners
* open fracture
* clinical signs of foot deformity
* previous foot trauma or surgery on the affected foot
* significant osteoarthritis or pre-existing ligamentous instability or pain in the affected foot
* unable to stand in the weight bearing position during the CT scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been diagnosed with unstable supination-external rotation type ankle fractures
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2016-02; Primary Completion 2017-02-02 (Actual); Study Completion 2017-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Marzo, MD, Principal Investigator — UBMB Orthopaedics & Sports Medicine
Locations (1):
- UBMD Orthopaedics & Sports Medicine, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ankle Fracture Cases: 9 patients with SER ankle fractures
Period: Overall Study
Arm/Group | Ankle Fracture Cases
Started (Enrolled in the study) | 9
Completed (Completed the study) | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Ankle Fracture Cases: 9 ankle fractures included in the study
Arm/Group | Ankle Fracture Cases
Number analyzed (Participants) | 9
Age, Continuous [Mean (Full Range); unit: years] | 50.3 [33 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 6

OUTCOME MEASURES:

1. Primary Outcome: Medial Clear Space Distance in the Ankle Joint
Description: measured on weight bearing CBCT
Time Frame: Baseline- single-day study
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Ankle Fracture Cases
Number analyzed (Participants) | 9
mm | 1.41 (0.41)

2. Secondary Outcome: Medial Clear Space on Gravity Stress Xray
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Ankle Fracture Cases
Number analyzed (Participants) | 9
mm | 5.82 (1.93)

3. Secondary Outcome: Medial Clear Space on Standard Xray
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Ankle Fracture Cases
Number analyzed (Participants) | 9
mm | 3.28 (1.63)

ADVERSE EVENTS:
Time Frame: not monitored beyond the study visit
Description: There is no risk of serious adverse events, including death, involved with this study.
Arm/Group | Ankle Fracture Cases
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-11): https://cdn.clinicaltrials.gov/large-docs/41/NCT02599441/Prot_SAP_000.pdf